CLINICAL TRIAL: NCT06214702
Title: Deregulated Serum Levels of Serpin C and Soluble Fms-like Tyrosine Kinase-1 Might Predict the Development of Preeclampsia in Normotensive Pregnant Women
Brief Title: Serpin C and Soluble Fms-like Tyrosine Kinase-1 Levels in Normotensive Pregnant Women May Predict the Development of Preeclampsia
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Omar K. Naser, lecturer of obstetrics and gynecology, Benha University
Other Study IDs: RC 7.1.2024
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with diastolic blood pressure (DBP) after the 20th GW up ≥140 or 90 mmHg without proteinuria.
  Interventions: Diagnostic Test: ELISA
- Control Group: Patients were normotensive at the 20th GW.
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — ELISA estimation of PLGF, sFlt-1 and Serpin C

SUMMARY:
Evaluation of the predictability of estimated levels of Serpin C, sFlt-1 and placental growth factor (PLGF) in blood samples obtained during the 1st trimester from normotensive pregnant women for identification of women liable to develop PE during the course of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive pregnant women had singleton fetus presenting during the 1st trimester
* free of exclusion criteria

Exclusion Criteria:

* Age
* Sex
* Hypertension

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients were having monthly follow-up of pregnancy and determination of BP measures, and estimation of the serum levels of the studied biomarkers.
  Patients who developed GHTN at the 20th GW were grouped as GHTN group and those who were normotensive at the 20th GW were considered as control.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Role of Biomarkers in detection of GHTN | 9 months
  The predictability of serum biomarkers' levels estimated at enrolment for the development of GHTN.

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, El- Qalyobia, Egypt